CLINICAL TRIAL: NCT04436224
Title: Hydromorphone for ICU-analgesia in Patients With Non-mechanical Ventilation: A Dose-exploration and Effectiveness Study
Brief Title: Hydromorphone for ICU-analgesia in Patients With Non-mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Zhenhua Zen, Associate Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nfyyicu002
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Hydromorphone; Analgesia; ICU
MeSH Terms: conditions — Agnosia | interventions — Hydromorphone; Fentanyl; Butorphanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hydromorphone (Experimental): NS 40ML+ hydromorphone(10mg , 2mg:2ml），IV-Pump，maintenance dose 0.50mg/h
  Interventions: Drug: Hydromorphone
- fentanyl (Active Comparator): NS 40ML+ fentanyl(0.5mg, 0.1mg:2ml），IV-Pump，maintenance dose 0.08-0.2mg/h
  Interventions: Drug: Fentanyl
- Butorphanol (Active Comparator): NS 40ML+ butorphanol(10mg, 1mg:1ml），IV-Pump，maintenance dose 0.7-10mg/kg/h
  Interventions: Drug: Butorphanol

INTERVENTIONS:
Drug: Hydromorphone — Intravenous analgesia using hydromorphone in ICU patients with non-mechanical ventilation(NS 40ML+ hydromorphone 10mg ，IV-Pump)
  Arms: hydromorphone
Drug: Fentanyl — Intravenous analgesia using fentanyl in ICU patients with non-mechanical ventilation(NS 40ML+ fentanyl 0.5mg, IV-Pump)
  Arms: fentanyl
Drug: Butorphanol — Intravenous analgesia using butorphanol in ICU patients with non-mechanical ventilation(NS 40ML+ butorphanol 10mg，IV-Pump)
  Arms: Butorphanol

SUMMARY:
Hydromorphone has a clear analgesic effect, and has few advantages in respiratory depression and gastrointestinal motility. The study will further explore the continuous pumping-dose of hydromorphone for ICU non-mechanical ventilation patients and monitor its effective plasma concentration as well as evaluates the safety and effectiveness of hydromorphone for ICU non-mechanical ventilation patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Non-mechanical ventilation patients with expected ICU stay time >24h
* People with moderate to severe pain who need immediate analgesic treatment (NRS ≥ 4 or BPS ≥ 5 points, CPOT ≥ 3);

Exclusion Criteria:

* pregnancy；
* can not get pain score from patients
* allergy to drugs
* ....

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
successful analgesic proportion | From date of using the intervention drugs until the date of leaving from icu, up to 28 days
  Proportion of patients in each group who reached the target analgesia score range

SECONDARY OUTCOMES:
Score | From date of using the intervention drugs until the date of stopping using intervention drugs, up to 28 days
  analgesia score, such as CPOT or NRS
dose of analgesics | From date of using the intervention drugs until the date of stopping using intervention drugs, up to 28 days
  total dose of analgesics during the study
Adverse event | From date of using the intervention drugs until the date of discharge or death from any cause, up to 60 days
  Adverse event during the study, including hypotension.et
ICU stay | from the date of entering icu until the date of leaving icu or death from any cause, up to 28 days.
  duration of stay in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Southern medical university Nanfang hospital, Guangzhou, China